CLINICAL TRIAL: NCT04352907
Title: Accuracy of Dexcom G6 Continuous Glucose Sensor in the Intensive Care Unit
Brief Title: Accuracy of CGM in the ICU, Compared to Standard of Care
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of British Columbia (Other)
Collaborators: DexCom, Inc. (Industry)
Responsible Party: Principal Investigator, David Thompson, Clinical Assistant Professor, University of British Columbia
Other Study IDs: H19-02392
Record Dates: First submitted 2020-04-15; First posted 2020-04-20 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2022-05

CONDITIONS: Diabetes
Keywords: insulin infusion; continuous glucose sensor
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

INTERVENTIONS:
Device: Continuous Glucose Sensor — Continuous glucose sensor results will be compared with arterial glucose samples

SUMMARY:
To determine the performance of the Dexcom CGM device in comparison to arterial glucose samples.

DETAILED DESCRIPTION:
The performance of the Dexcom continuous glucose sensor will be compared with the current standard of care which is arterial glucose samples analyzed on a glucose meter. Subjects will be ICU patients receiving intravenous insulin infusions.

ELIGIBILITY:
Inclusion Criteria:

* minimum age 18 years
* anticipated to be on an insulin infusion for 3-7 consecutive days
* 10 of these subjects will be on vasopressors who will be receiving large volume fluid resuscitation

Exclusion Criteria:

* subjects not on insulin infusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects in the Intensive Care Unit
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2020-11-06 (Actual); Primary Completion 2022-09 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Continous Glucose Sensor values (CGM) | 3 to 7 consecutive days
  CGM will be compared with arterial glucose values

SECONDARY OUTCOMES:
Vasopressor Use | 3 to 7 consecutive days
  10 of the 20 subjects will be on vasopressors and large volume fluid resuscitation

CONTACTS AND LOCATIONS:
Locations (1):
- Vancouver General Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No